CLINICAL TRIAL: NCT01481025
Title: Phase 3 Study - Efficacy and Tolerance for the Mixture of Dry Extracts Black Cohosh and Saint John's Worth Versus Isolated Black Cohosh Extract for the Climacteric Symptoms' Control
Brief Title: Efficacy and Safety for Cimicifuga/Hypericum Product
Acronym: CH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Phytopharm Consulting Brazil (Network)
Collaborators: Herbarium Laboratorio Botanico Ltda (Industry); Complexo Hospitalar Santa Casa de Misericordia de Porto alegre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cimicifuga/Herbarium
Record Dates: First submitted 2011-11-25; First posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Perimenopausal Disorder
Keywords: Climacteric; Depression; Herbal treatment
MeSH Terms: conditions — Depression | interventions — black cohosh root extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cimicifuga+Hiperico (Experimental): 80 + 450 mg / tablet
  Interventions: Drug: Cimicifuga + Hiperico
- Cimicifuga Herbarium (Active Comparator): 80 mg / caps
  Interventions: Drug: Cimicifuga Herbarium
- Aplause® (Active Comparator): 20 mg / tablet
  Interventions: Drug: Aplause®

INTERVENTIONS:
Drug: Cimicifuga + Hiperico — 1 tablet, 80+450mg/tablet, twice a day for 1-3 months
  1 tablet, 80+450mg/tablet, once a day for 3-6 months
  Arms: Cimicifuga+Hiperico
Drug: Cimicifuga Herbarium — 2 caps, 80mg/caps, once a day for 1-3 months
  1 caps, 80mg/caps, once a day for 3-6 months
  Arms: Cimicifuga Herbarium
Drug: Aplause® — 4 tablets, 20mg/tablet, twice a day for 1-3 months 2 tablets, 20mg/tablet, twice a day for 3-6 months
  Arms: Aplause®

SUMMARY:
Climacteric Complains bring to women many problems for living a normal life - hot flashes, irritation are 2 of many problems and the mixture of those 2 plant extract must bring a new horizon for this part of time.

DETAILED DESCRIPTION:
2 herbal extracts used in general alone will be running together for the best climacteric women on quality of life.

The investigators will test the mixture already in the market as GynoPlus and RemifeminPlus, but as each extract has its own particularities the investigators will try CIM/HIP as a unique formulation versus Clifemin® as control and Aplause® as comparator.

This protocol was performed for the best of our volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Climacteric women 45-60 years old - pre and postmenopausal
* Climacteric complains for at least 3 months
* No treatments for at least 2 months
* MRS score 0.4 or more for at least 3 items
* Hamilton's Scale score from 15-23

Exclusion Criteria:

* Hormon Therapy or any other for the last 3 months
* Antidepressive and Hypnotic medication for the last 3 months
* Sever illness (cardiac, hepatic, renal, digestive or metabolic) or TSH alteration
* History for allergies and hipersensitivity to any component of the drugs formulations
* No knowledge for reading or writing
* Suicide risk

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-06 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Menopause Rating Scale | 8 months
  Climacteric Symptoms Evaluation - "MRS - Menopause Rating Scale*

SECONDARY OUTCOMES:
Hamilton's Depression Scale | 8 months
  Questionair for Depression Symptoms
WHOQOL | 8 months
  Starting Point (T-2) and Ending Point (T6)
Health Numbers | 8 months (T-2 to T6)
  Starting Point (T0, T1, T3 and T6)

CONTACTS AND LOCATIONS:
Overall Officials: Karla F Deud José, Pharm PhD, Study Chair — Phytopharm Consulting Brazil - karla@phytopharm.com.br; Carla Vanin, MD MSc PhD, Principal Investigator — Federal University of Health Science of Porto Alegre; Raquel P Dibi, MD MSc, Principal Investigator — Irmandade Santa Casa de Misericórdia de Porto Alegre
Locations (1):
- ISCMPA's Gynecology Ambulatory, Porto Alegre, Rio Grande do Sul, Brazil